CLINICAL TRIAL: NCT01857128
Title: A Prospective Randomized Open-Label Study Examining the Efficacy of Drawtex® Hydroconductive Wound Dressing and Negative Pressure Wound Therapy in Pilonidal Cystectomy Wounds Healing by Secondary Intention - A Pilot Study
Brief Title: Pilonidal Disease Wound Healing Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael P. McNally, Principal Investigator, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 382094-2
Record Dates: First submitted 2013-05-07; First posted 2013-05-20 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Pilonidal Disease
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drawtex Hydroconductive Dressing (Experimental): Gauze-like dressing placed onto wound
  Interventions: Device: Drawtex dressing
- Negative Pressure Wound Therapy (Active Comparator): Usual care including vacuum and canister
  Interventions: Device: Negative Pressure Wound Therapy

INTERVENTIONS:
Device: Drawtex dressing
  Arms: Drawtex Hydroconductive Dressing
Device: Negative Pressure Wound Therapy
  Arms: Negative Pressure Wound Therapy

SUMMARY:
The purpose of the study is to learn about the best way to treat pilonidal cyst wounds and learn which type of bandage (or dressing) can help the wound heal faster after having surgery.

DETAILED DESCRIPTION:
This pilot study is a prospective randomized open-label study examining the efficacy of Drawtex® Hydroconductive wound dressing and negative pressure wound therapy(NPWT) in pilonidal cystectomy wound healing by secondary intention.

Pilonidal disease has a significant impact on the active duty demographic and the treatments for this disease result in a substantial cost to the military in both duty days lost and for the medical care provided. This study examines Negative Pressure Wound Therapy (NPWT) and the Drawtex® Hydroconductive Dressing for the treatment of surgical wounds resulting from limited excision of pilonidal disease. This clinical trial is a prospective, randomized open label examination of two standard wound therapy modalities with the goal of determining which treatment promotes the most rapid wound healing by secondary intention. Secondary goals include determining which treatment is most cost effective and is most acceptable to patients.

Active duty, retired, and dependent adults (age 18-60 years) who are scheduled to undergo limited surgical cyst excision will be recruited from patients who are referred to the General Surgery Department at Walter Reed National Military Medical Center (WRNMMC). Health care providers in the General Surgery Department will be informed about the study and requested to refer appropriate patients to the study Investigators for evaluation and potential inclusion in the study. The informed consent process will occur at WRNMMC, General Surgery Clinic during the pre-operative clinic visit(s). If the patient consents to screening for inclusion in the study, then they will be assigned a subject number and randomly assigned to a study arm, either NPWT or Drawtex®, preoperatively. The subject will then undergo a limited excision of the pilonidal cyst. If the resulting wound post-surgery meets enrollment criteria, then the subject will be enrolled in the study. At this point, the randomization arm will be revealed either NPWT or Drawtex® dressing. Wound care will be done at the wound care clinic two times a week (biweekly) for approximately 4 weeks or until there is 75% epithelialization, and then on a weekly and then on a monthly basis until 100% epithelialization of the wound or 270 days of follow up are reached. Wound healing progress will be evaluated objectively using a digital planimetry analysis system and blinded evaluators. Secondary objectives include adverse events, bacterial load, expression of inflammatory markers, cost to military and patient satisfaction assessments,

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or non-lactating female age 18 to 60 years inclusive.
2. Diagnosis of pilonidal disease with cyst requiring surgery, with undermining to remove the cyst and requiring limited excision with healing by secondary intension.
3. Presence of chronic symptomatic pilonidal disease defined as at least one pilonidal sinus and a history of at least two acute pilonidal abscesses or persistent symptoms altering patient's quality of life.
4. Military active duty members need a supervisor signed memorandum to participate (Active Duty Supervisor's Approval Memo).
5. Understands the purpose and risks of study by scoring 80% or higher on knowledge assessment test.
6. Available and willing to participate for the duration of the study (approximately 30-270 days maximum depending on time to wound healing).
7. Available and willing to provide written informed consent.
8. Able and willing to follow instructions as per protocol.
9. Available for all visits as per protocol. Post Surgery Study Enrollment Criteria
10. Post-surgical wound measurement (length x width x depth):

(cm x 1.5 cm x 1.5 cm)greater than or equal to 3 cm in length, greater than or equal to 1.5 cm in width, and greater than or equal to1.5 cm in depth.

Rationale: satisfies the minimum size wound that NPWT may be employed.

Exclusion Criteria:

1. Does not meet all inclusion criteria.
2. Pregnant (by history or as ascertained by pregnancy test) or lactating female Rationale: immune modulation and potential for altered healing trajectory as well as operative risk to fetus for elective procedure.
3. Known HIV infection.
4. Known immunodeficiency or currently receiving immunosuppressive therapy (inhaled and topical steroids are allowed).
5. Autoimmune disease (clinical, preexisting anti-dsDNA antibodies 30 IU, or positive ANA ELISA with a titer greater than 1:80 on pre-operative screening) Exclusionary medical histories will include the following diagnoses: systemic lupus erythematosus, rheumatoid arthritis, mixed connective tissue disease, progressive systemic sclerosis, Sjogren's syndrome, polymyositis/ dermatomyositis, and vasculitis Rationale: potential for altered wound healing.
6. Acute or chronic, clinically significant cardiac, pulmonary, hepatic, or renal abnormality, as determined by physical examination or basic laboratory screening performed at pre-operative evaluation.
7. Known documented history of diabetes mellitus.
8. Non-ambulatory or limited mobility. Rationale: non ambulatory patients may have altered wound healing in the sacral area due to constant pressure from positioning.
9. History of current tobacco use: defined as cigarette smoking greater than or equal to one half pack (10 cigarettes) per day:

   Rationale: confounding factor prolonging wound healing.
10. Complex pilonidal disease determined by the surgeon to require a procedure other than the study procedure for appropriate treatment of the disease.
11. Acute pilonidal abscess or infection within 6 weeks of planned operative date.
12. Concerns for arterial bleeding or cancer in the wound bed or in the vicinity of the dressing.
13. Any other significant finding which, in the opinion of the investigator, would increase the subject's risk of having an adverse outcome from participating in this protocol.
14. Lack of or unwillingness to provide/sign informed consent. Post Surgery Exclusion Study Criteria
15. Post-surgical wound measurement restrictions (enth x width x depth):

(0 cm x 10 cm x 6 cm)greater than or equal to 10 cm in length, greater than or equal to 10 cm in width OR greater than or equal to 6 cm in depth. If bone is visible or exposed, the subject must be excluded.

Rationale: large wounds are deemed complex and wounds with exposed or visible bone require antibiotic therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to wound healing | Up to 270 days or 9 months
  Time (days) to 100% epithelialization of the wound bed will be evaluated using digitized planimetry in a random manner by two independent evaluators blinded to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P McNally, M.D., Principal Investigator — Department of General Surgery
Locations (1):
- Walter Reed National Military Medical Center -Dept of General Surgery, Bethesda, Maryland, United States